CLINICAL TRIAL: NCT00832351
Title: Effect of Immediate Mobilisation After Stroke on Mortality, Morbidity and Functional Outcome
Brief Title: Akershus Early Mobilisation in Stroke Study
Acronym: AKEMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Antje Sundseth, MD, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.2006.322 (REK); 04/01666-22 (NSD)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Stroke
Keywords: Stroke; Brain infarction; Intracerebral hemorrhage; Early Mobilisation
MeSH Terms: conditions — Stroke; Brain Infarction; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Early mobilisation within 24 hours after admittance to hospital
  Interventions: Procedure: Mobilisation
- 2 (No Intervention): Mobilisation after 24 but within 48 hours from admittance to hospital

INTERVENTIONS:
Procedure: Mobilisation — Mobilisation
  Arms: 1

SUMMARY:
Treatment in stroke units compared with treatment in general medical wards reduces the odds of being dead or disabled. Little is known about which components of acute stroke care that is responsible for this benefit.

Early mobilisation is one of the features of stroke unit care. In Scandinavia, any intervention aimed to reduce the time to the first out of bed episode has been focused in order to prevent complications.

However, therapeutic interventions for cerebral revascularisation and a more intensive unit approach for observation may postpone mobilisation. The aim of the present study is to identify whether early mobilisation (< 24 hours after admittance to hospital)reduce disability and mortality compared with mobilisation after 24 hours.

The study is a prospective, randomised controlled study with blinded assessment at the end of follow up. Patients admitted to the Stroke Unit, Akershus University Hospital less than 24 hours after stroke during 2009 - 2011 are screened for recruitment. Patients are randomly assigned to either mobilisation out of bed within 24 hours from admittance to hospital or mobilisation after 24 hours. Except early contra late mobilisation all patients receive standard stroke unit care.

Patients with modified Rankin Scale 0 and 1, patients with a secondary intracerebral hemorrhage, patients receiving thrombolysis or patients requiring palliative care are excluded.

All patients are assessed at admittance, discharge and 3 months poststroke. Investigations at admittance include standard blood sample, CT/MRI scan, EKG and ultrasound of carotid arteries.

Main outcome is mortality and disability 3 months poststroke. Secondary outcome measures are neurological deficits (NIH), morbidity, complications, cognitive function reflected by Mini Mental State Examination and emotional function (Hospital Anxiety and Depression scale) .

Results from this study may add important knowledge about how and when to start mobilisation of patients with acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the Department of Neurology, Akershus University Hospital, with acute stroke (ischemic or hemorrhagic)

Exclusion Criteria:

* admitted to hospital more than 24 hours after stroke onset
* mRS 0 and 1
* mRS 5
* patients requiring palliative care
* secondary/traumatic intracerebral hemorrhage
* pregnancy
* i.v./i.a. thrombolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Effect of early mobilisation after stroke (< 24 hours after admittance to hospital) on mortality, morbidity and functional outcome | 3 month

SECONDARY OUTCOMES:
Neurological deficits | 3 month
  NIHSS
Morbidity | 3 month
Complications | 3 month
Cognitive function | 3 month
  MMSE
Emotional function | 3 month
  HAD

CONTACTS AND LOCATIONS:
Overall Officials: Ole Morten Rønning, MD, PhD, Study Chair — Department of Neurology, Akershus University Hospital
Locations (1):
- Department of Neurology, Akershus University Hospital, Lørenskog, Akershus, Norway